CLINICAL TRIAL: NCT01909947
Title: Prediction of Extubation Readiness in Extreme Preterm Infants by the Automated Analysis of CardioRespiratory Behavior: the APEX Study
Brief Title: Prediction of Extubation Readiness in Extreme Preterm Infants by the Automated Analysis of CardioRespiratory Behavior
Status: Completed | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Wayne State University (Other); Brown University (Other)
Responsible Party: Principal Investigator, Guilherme Sant'Anna, MD, Associate Professor of Pediatrics, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: APEX 01; 288299 (Other Grant/Funding Number: CIHR); 12-387-PED (Other: MUHC)
Record Dates: First submitted 2013-07-17; First posted 2013-07-29 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Prediction of Extubation Readiness
Keywords: Respiratory rate variability; Heart rate variability; Extubation readiness; Extubation failure; Clinical predictors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intubated extreme preterm infants: Infants with a birth weight ≤ 1250 grams and requiring endotracheal tube and mechanical ventilation
  Interventions: Other: Cardiorespiratory signal acquisition

INTERVENTIONS:
Other: Cardiorespiratory signal acquisition — Cardiorespiratory signals will measure heart rate (using electrocardiography), chest and abdominal movements (using respiratory inductance plethysmography) and oxygen saturation (using pulse oximetry). Data will be acquired during 2 recording periods:
  1. A 60-minute period while the infant receives any mode of conventional mechanical ventilation
  2. A 5-minute period prior to extubation while the mode of ventilation is switched to endotracheal tube CPAP (Continuous Positive Airway Pressure), so that the respiratory pattern will be controlled by the infant

SUMMARY:
The investigators hypothesize that machine learning methods using a combination of novel, quantitative measures of cardio-respiratory variability can accurately predict the optimal time to extubate extreme preterm infants. In this multicenter prospective study, cardiorespiratory signals will be recorded from 250 extreme preterm infants who are eligible for extubation. Automated signal analysis algorithms will compute a variety of metrics for each infant describing the cardiorespiratory state. Machine learning methods will then be used to find the optimal combination of these statistical measures and clinical features that provide the best overall predictor of extubation readiness. Finally, investigators will develop an Automated system for Prediction of EXtubation (APEX) that will integrate the software for data acquisition, signal analysis, and outcome prediction into a single application suitable for use by medical personnel in the Neonatal Intensive Care Unit (NICU). The performance of APEX will later be clinically validated in 50 additional infants prospectively.

DETAILED DESCRIPTION:
At birth, extreme preterm infants (≤28 weeks) have inconsistent respiratory drive, airway instability, surfactant deficiency and immature lungs that frequently result in respiratory failure. Management of these infants is difficult and most will require endotracheal intubation and mechanical ventilation (ETT-MV) within the first days of life to survive. ETT-MV is an invasive therapy that is associated with adverse clinical outcomes including ventilator-associated pneumonia, impaired neurodevelopment, and increased mortality. Consequently, clinicians try to remove ETT-MV as quickly as possible. However, 25 to 35% of these extubation attempts will fail and infants will require reintubation, an intervention that is also associated with increased morbidity and mortality. Therefore physicians must determine the optimal time for extubation which minimizes the duration of ETT-MV and maximizes the chances of success. A variety of objective measures have been proposed to assist with this decision but none has proven to be useful clinically. Investigators from this group have recently explored the predictive power of indices of autonomic nervous system function based on measurements of heart rate (HRV) and respiratory variability (RV). The use of sophisticated, automated algorithms to analyze those cardiorespiratory signals have shown some promising preliminary results in predicting which infants can be extubated successfully.

ELIGIBILITY:
Inclusion Criteria:

* All infants admitted to the NICU with a birth weight ≤ 1250 grams AND
* Need for endotracheal tube mechanical ventilation

Exclusion Criteria:

* Infants with major congenital anomalies
* Infants with congenital heart disease and cardiac arrhythmias
* Infants receiving vasopressor or sedative drugs at the time of extubation
* Infants extubated directly from high frequency ventilation
* Infants extubated to room air, oxyhood or low-flow nasal cannula

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Extreme preterm infants who are requiring endotracheal tube mechanical ventilation (ETT-MV).
Sampling Method: Non-Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Extubation Failure | Within 72 hours of extubation
  Infants will be considered to have failed extubation if they meet one or more of the following criteria within 72 hours of extubation:
  1. Fraction of inspired oxygen (FiO2) > 0.5 in order to maintain oxygen saturation (SpO2) > 88% or PaO2 > 45 mmHg (for 2 consecutive hours)
  2. PaCO2 > 55-60 mmHg with a pH < 7.25 in two consecutive blood gases done 1-2 hours apart
  3. 1 episode of apnea requiring positive pressure ventilation with bag and mask
  4. Multiple episodes of apnea (≥ 6 episodes / 6 hours).

SECONDARY OUTCOMES:
The need for reintubation within 72h of the first planned extubation | Within 72 hours of extubation
  The decision to re-intubate will be made by the responsible physician, who may not always follow the guidelines stated in the primary objective. Therefore, reintubation will be assessed as a secondary outcome.
The need for reintubation | Anytime from the first planned extubation until discharge from the neonatal intensive care unit
  Infants will be prospectively followed from birth until discharge from the NICU. Therefore, infants who require reintubation at any time point from the first planned extubation until discharge from the neonatal intensive care unit will be documented

OTHER OUTCOMES:
Total duration of ETT-MV | Participants will be followed for the duration of hospital stay, an expected average of 10 weeks
  Total duration (in days) of endotracheal tube mechanical ventilation from the time of birth until discharge from the hospital
Intraventricular hemorrhage | Participants will be followed for the duration of hospital stay, an expected average of 10 weeks
  Presence of Intraventricular Hemorrhage (IVH) from time of birth until discharge from the hospital. If IVH is present, the grade of the hemorrhage will be specified (as per Volpe's classification)
Patent Ductus Arteriosus | Participants will be followed for the duration of hospital stay, an expected average of 10 weeks
  Presence of a Patent Ductus Arteriosus (PDA) from the time of birth until discharge from hospital. If present, the therapeutic measures taken for closing the PDA (medical or surgical) will also be specified.
Oxygen supplementation at 28 days of life | This outcome will be assessed when participants have 28 days of life
  The need for any oxygen supplementation at 28 days of life
Bronchopulmonary Dysplasia | This outcome will be assessed when participants are 36 weeks post-conceptual age
  The presence of Bronchopulmonary Dysplasia (BPD) will be assessed at 36 weeks Post Conceptual Age (PCA) and classified as mild, moderate or severe.
  * Mild BPD: oxygen supplementation at 28 days of life but none at 36 weeks PCA
  * Moderate BPD: FiO2 requirements of less than 0.3 at 36 weeks PCA
  * Severe BPD: FiO2 requirements over 0.3 or CPAP or mechanical ventilation at 36 weeks PCA
Retinopathy of Prematurity | This outcome will be assessed at the time of the first eye exam (approximately 31 weeks PCA) until the final eye exam prior to hospital discharge
  Participants will be assessed for the presence or absence of Retinopathy of Prematurity (ROP)
Necrotizing Enterocolitis | Participants will be followed for the duration of hospital stay, an expected average of 10 weeks
  Participants will be assessed for the presence or absence of Necrotizing Enterocolitis (NEC) throughout the course of their hospitalization. NEC will be classified according to Bell's modified staging criteria.
Death | Participants will be followed for the duration of hospital stay in the NICU, an expected average of 10 weeks
  Death occuring anytime during the hospitalization course in the NICU.

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme M Sant'Anna, MD, Study Chair — McGill University; Guilherme M Sant'Anna, MD, Principal Investigator — McGill University; Robert E Kearney, PhD, Principal Investigator — McGill University; Wissam Shalish, MD, Principal Investigator — McGill University; Karen A Brown, MD, Principal Investigator — McGill University; Doina Precup, Principal Investigator — McGill University; Sanjay Chawla, MD, Principal Investigator — Wayne State University; Martin Keszler, MD, Principal Investigator — Brown University
Locations (5):
- United States (2):
  - Wayne State University, Detroit, Michigan
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
- Canada (3):
  - Royal Victoria Hospital, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Alarcon-Martinez T, Latremouille S, Kovacs L, Kearney RE, Sant'Anna GM, Shalish W. Clinical usefulness of reintubation criteria in extremely preterm infants: a cohort study. Arch Dis Child Fetal Neonatal Ed. 2023 Nov;108(6):643-648. doi: 10.1136/archdischild-2022-325245. Epub 2023 May 16. PMID 37193586
- [Derived] Shalish W, Kanbar LJ, Rao S, Robles-Rubio CA, Kovacs L, Chawla S, Keszler M, Precup D, Brown K, Kearney RE, Sant'Anna GM. Prediction of Extubation readiness in extremely preterm infants by the automated analysis of cardiorespiratory behavior: study protocol. BMC Pediatr. 2017 Jul 17;17(1):167. doi: 10.1186/s12887-017-0911-z. PMID 28716018